CLINICAL TRIAL: NCT06536296
Title: The Impact of Music Medicine on Preterm Brain Development and Behavior - A Two-Center Randomized Controlled Trial "The Lullaby Study"
Brief Title: The Impact of Music Medicine on Preterm Brain Development and Behavior
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Yale New Haven Health System Center for Healthcare Solutions (Other)
Responsible Party: Principal Investigator, Carmina Erdei, MD, Neonatologist, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2024P001561
Record Dates: First submitted 2024-07-10; First posted 2024-08-02 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Infant Development; Language Development; Prematurity; Stress
Keywords: Preterm; Neurodevelopment; Music-based Intervention
MeSH Terms: conditions — Premature Birth | interventions — Music Therapy; Standard of Care

STUDY DESIGN:
Intervention Model Description: The eligible participants in both institutions will be consecutively approached to enroll in the study. Once informed consent has been obtained, each participant will be randomly assigned to one of the three study groups: M (music), MPV (music with parent voice), or SC (standard care), with 81 infants per each group. We designed the MBI in collaboration with board certified music therapists (MT) at the two institutions. While MBI recordings will be obtained at each NICU timepoint for each infant (with both M and MPV; SC group will wear headphones open to environmental sounds, as a control group), each infant will only listen to one of the three types of recordings according to their group assignment.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: We will utilize infant-adapted headphones to deliver the intervention in a blinded fashion. The research team (investigators and outcome assessors) will remain blinded to the type of recording delivered for each infant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music (Experimental): We will create three recordings with increasing complexity for each infant. For each infant developmental stage (32, 34, 36+ weeks PMA), Music Therapists (MTs) in both units will present parents with a curated list of 8-10 musically comparable, familiar lullabies to select from. Songs will be available in different languages reflective of patient diversity, with rhythm, tempo, pitch range/ change, instrumentation, melody, harmony selected drawing on available evidence, including BWH NICU pilot data. Timing: MBI to be administered after regular NICU "care and feeding" times, which are typically considered stressful times for infants. The goal of the intervention will be to provide a calming and relaxing experience to the infant as they "settle" back to sleep after handling times. Music delivery will occur via infant-adapted headphones to facilitate blinding.
  Interventions: Other: Music
- Music and parent voice (Experimental): The selected lullabies will be pre-recorded by the MT as described above to include a guitar accompaniment track, and a separate vocal track with the MT singing along, in two separate keys to allow variation for parent voice range and comfort. Parents will be invited to sing along with the recorded track of MT singing, and MT will later remove the MT-voice recording track so only the parent voice will be heard with the guitar in the final recording. Timing: MBI to be administered after regular NICU "care and feeding" times, which are typically considered stressful times for infants. The goal of the intervention will be to provide a calming and relaxing experience to the infant as they "settle" back to sleep after handling times. Music delivery will occur via infant-adapted headphones to facilitate blinding.
  Interventions: Other: Music and parent voice
- Reference/ Standard of care (Active Comparator): These are infants recruited in the study who will receive the unit standard of care. They will be listening to the NICU ambient noise via infant-adapted headphones but will not receive any music intervention.
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Music — Arm 1: Music only
  Other Names: Arm 1: Music
  Arms: Music
Other: Music and parent voice — Arm 2: Music and parent voice
  Other Names: Arm 2: Music and parent voice
  Arms: Music and parent voice
Other: Standard Care — Standard Care
  Other Names: Arm 3: Standard Care
  Arms: Reference/ Standard of care

SUMMARY:
The investigators are conducting a two-site randomized control trial with the aim of defining the impact of music (M) without or with parent voice (MPV) on very preterm infants' acute and cumulative stress, intranetwork connectivity on term brain MRI, and language and other neurodevelopmental outcomes at two years corrected age. This is based on the hypothesis that infants in MPV arm are expected to experience the greatest benefit compared with infants receiving standard care.

DETAILED DESCRIPTION:
Preterm birth remains the leading cause of death for children under five. For survivors, it also accounts for high morbidity and substantial physical, psychosocial, emotional, and financial burden for individuals, families, and communities. The impairments span over multiple domains, with language difficulties affecting about half of surviving children. Evidence indicates that preterm birth has significant impacts on long-term functioning, yet primary prevention of preterm birth is presently not feasible. It is therefore imperative to prioritize early interventions to mitigate these adverse long-term effects on child and family outcomes.

Very preterm (VP) infants, i.e., those born below 32 weeks gestational age (GA) typically spend 2-4 months hospitalized in the Neonatal Intensive Care Unit (NICU) before reaching term-equivalent age (TEA). During this time, the preterm brain nearly quadruples in volume and is highly sensitive to both positive and negative environmental experiences. Yet, during this period, VP infants must also receive life-saving intensive medical care in the sensory-atypical environment of the NICU. From an auditory perspective, this atypical environment comprises loud equipment sounds at volumes far exceeding recommended levels, silence, and a paucity of human interaction. One domain of neurosensory experience is the auditory environment, comprised predominantly of non-meaningful, high-frequency/ high decibel equipment sounds, and silence. The deprivation of VP infants from enriching auditory experiences (parental voice, infant-directed language) combined with the constant influx of high frequency/high decibel sounds (alarms and electronic noise) can induce chronic stress and negatively impact auditory and other areas of cortical development.

For preterm infants who have not yet reached term-equivalent age (TEA), the NICU hospitalization is a critical window for developmental adaptability to experience during a highly sensitive period of brain development. There are two key pathways whereby music and voice therapy in the VP infant are thought to have benefit - stress reduction and auditory enrichment. Recent work indicates that music therapy may reduce the immediate stress experienced by VP infants, with evidence emerging on its impact to improve neurodevelopmental outcomes. Prior studies have been limited due to small size, variability of music exposures, inconsistent study design and outcome measures. Further, most studies explored exposure-outcome associations, without mechanistic investigation. One study showed improved white matter maturation in acoustic radiations, larger amygdala volumes, and enhanced functional connectivity brain magnetic resonance imaging (MRI) after early music exposures. These suggests that early music exposure may enhance auditory cortex development and reduce stress (amygdala) in VP infants.

While small studies inform these hypotheses, a large, randomized trial is necessary to test them more rigorously. Our own center's pilot study demonstrated that a music condition with low, repetitive, and rhythmically consistent entrainment stimulus was associated with improved physiologic state after the exposure. Based on these data, the investigators plan to further develop an individualized intervention encompassing evidence-based musical elements onto which parental voice will be carefully layered. The aim of this proposal is to conduct a randomized trial to determine the effects of a protocolized music-based intervention (MBI) with and without parental voice on stress reduction, early brain structure and function, and neurodevelopmental outcomes.

The investigators propose to address this knowledge gap in a large, two-center randomized controlled trial (RCT), employing a novel MBI tailored based on available preliminary data and inclusive of musical and non-musical elements to facilitate parent engagement, with comprehensive evaluation of relevant clinical, neuroimaging, and neurodevelopmental outcomes of VP infants up to two years of age. The impact of this work will be two-fold: this proposal will 1) generate rigorous evidence to specifically support the integration of music medicine as a therapeutic approach for VP infants in the NICU, and 2) strengthen the evidence base for neurosensory interventions for hospitalized infants, which will shift the framework of care in the NICU by leveraging developmental care interventions to optimize the outcomes of VP infants.

ELIGIBILITY:
Inclusion Criteria:

* Very preterm infants born between 24+0 and 30+6 weeks' gestational age (GA) from 2 level III NICUs (Brigham and Women's Hospital, Boston, MA and Yale New Haven, CT)
* Infants who are medically stable per the clinical care team

Exclusion Criteria:

* Infants with major genetic or congenital anomalies known to be associated with developmental delay
* Infants with severe brain injury (such as intraparenchymal hemorrhage, severe white matter injury)
* Infants who are severely ill infants for whom MBI is not feasible
* Infants of parents who cannot complete questionnaires in English or Spanish.

Ages: 24 Weeks to 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 243 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2030-08-30 (Estimated); Study Completion 2031-03-01 (Estimated)

PRIMARY OUTCOMES:
Bayley-4 language performance (SA3 primary outcome) | 2 years corrected age
  Study patients Language performance measured on the Bayley-4 at 2 years corrected age
Amygdala volume on MRI (SA1a, primary outcome) | At term-equivalent (~ 3 months of age), 37-41 weeks postmenstrual age (PMA)
  Amygdala volume as a proxy of cumulative stress measured on term-equivalent brain MRI
Intranetwork connectivity in Salience and Language networks (SA2a, primary outcome) | Term-equivalent (~ 3 months of age), 37-41 weeks postmenstrual age (PMA)
  We will measure the intranetwork connectivity in Salience and Language networks in infants exposed to music and music with parent voice compared those in SC arm at term-equivalent

SECONDARY OUTCOMES:
Infant physiology - oxygen saturation | From enrollment to term-equivalent 37-41 weeks PMA
  We will record infant physiologic vital signs (i.e. oxygen saturation) from infants' bedside monitor around each study intervention
Infant physiology - respiratory rate | From enrollment to term-equivalent 37-41 weeks PMA
  We will record infant physiologic vital signs (i.e. respiratory rate) from infants' bedside monitor around each study intervention
Infant physiology - heart Rate | From enrollment to term-equivalent 37-41 weeks PMA
  We will record infant physiologic vital signs (i.e. heart rate) from infants' bedside monitor around each study intervention
Telomere length | At enrollment and term-equivalent 37-41 weeks PMA
  Assess infant premature aging at term-equivalent by measurement of telomere length on blood samples
Neurodevelopmental assessment - cognitive outcomes | 2 years corrected age
  Study patients' cognitive performance measured on the Bayley-4 assessment at 2 years corrected age
Neurodevelopmental assessment - motor outcomes | 2 years corrected age
  Study patients' motor performance measured on the Bayley-4 assessment at 2 years corrected age
Neurodevelopmental assessment - child behavior outcomes | 2 years corrected age
  Study patients' behavioral performance measured on the Child Behavior Checklist at 2 years corrected age
Brain development | Term-equivalent age - 37-41 weeks PMA
  Brain development and injury classified using the established Kidokoro scoring system applied to term-equivalent brain MRI
Parent stress | From term-equivalent age to 2 years corrected age
  Assessment of parent stress (Parental Stressor Scale) using a standardized survey of families of study infants
Parent anxiety and depression | From term-equivalent age to 2 years corrected age
  Assessment of parent anxiety and depression (Hospital Anxiety and Depression Scale) using one standardized survey that provides a combined score
Infant Neurobehavior | Term-equivalent 37-41 weeks PMA
  We will assess infant neurobehavior using the Hammersmith Neonatal Neurological Examination at term-equivalent age 37-41 weeks PMA

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Yale New Haven Hospital, New Haven, Connecticut
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided